CLINICAL TRIAL: NCT01264432
Title: A Phase I Study of Veliparib (ABT-888) in Combination With Low-Dose Fractionated Whole Abdominal Radiation Therapy (LDFWAR) in Patients With Advanced Solid Malignancies With Peritoneal Carcinomatosis With Two Additional Dose Levels in Patients With Epithelial Ovarian, Fallopian or Primary Peritoneal Cancers and Intra-Abdominal Disease
Brief Title: Veliparib and Radiation Therapy in Treating Patients With Advanced Solid Malignancies With Peritoneal Carcinomatosis, Epithelial Ovarian, Fallopian, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02913; NCI-2012-02913 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NA_00043143; J1097; NA_00043143, J1097; CDR0000691881; 8813 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); 8813 (Other: CTEP); P30CA006973 (NIH); U01CA132123 (NIH); U01CA070095 (NIH); UM1CA186644 (NIH); UM1CA186691 (NIH)
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Adult Solid Neoplasm; Peritoneal Carcinomatosis; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Peritoneal Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Radiotherapy; Radiation; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (veliparib, LDRWAR) (Experimental): Patients receive veliparib PO BID on days 1-21 (days 5-21 of course 1). Patients undergo LDFWAR in BID on days 1 and 5 of weeks 1-3. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Veliparib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo LDFWAR
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Veliparib — Given PO
  Other Names: ABT-888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I trial studies the side effects and best dose of veliparib when given together with radiation therapy in treating patients with advanced solid malignancies (abnormal cells divide without control and can invade nearby tissues) with peritoneal carcinomatosis, epithelial ovarian, fallopian, or primary peritoneal cancer. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x rays to kill tumor cells. Giving veliparib with radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerable dose of veliparib in combination with low-dose fractionated whole abdominal radiation therapy (LDFWAR) in patients with peritoneal carcinomatosis from advanced solid malignancies. At dose levels 5 and 6: to determine the maximum tolerable dose of veliparib in combination with LDFWAR in patients with epithelial ovarian, fallopian or primary peritoneal cancers with intraabdominal disease.

II. Determine the safety and toxicity of the combination of veliparib in conjunction with LDFWAR in patients with peritoneal carcinomatosis from advanced solid malignancies; at dose levels 5 and 6: to determine the safety and toxicity of veliparib in combination with LDFWAR in patients with epithelial ovarian, fallopian or primary peritoneal cancers with intraabdominal disease.

SECONDARY OBJECTIVES:

I. Assess clinical activity of veliparib plus LDFWAR in patients with peritoneal carcinomatosis from advanced solid malignancies as assessed by response rate by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. At dose levels 5 and 6: to assess the clinical activity of veliparib plus LDFWAR in patients with epithelial ovarian, fallopian or primary peritoneal cancer and intraabdominal disease as assessed by response rate by RECIST 1.1 criteria.

II. Evaluate if microsatellite instability or baseline levels of various deoxyribonucleic acid (DNA) repair proteins (excision repair cross-complementing 1 [ERCC1], x-ray repair complementing defective repair in Chinese hamster cells 1 [XRCC1], breast cancer 1, early onset [BRCA1], breast cancer 2, early onset [BRCA2], poly [adenosine diphosphate (ADP)-ribosyl]ation [PAR]) correlate with clinical activity of this regimen.

III. Evaluate changes in quality of life for patients treated with this regimen by serial measurements using the Quality of Life Questionnaire Core-30 (QLQC-30) standardized questionnaire.

OUTLINE: This is a dose-escalation study of veliparib.

Patients receive veliparib orally (PO) twice daily (BID) on days 1-21 (days 5-21 of course 1). Patients undergo LDFWAR in BID on days 1 and 5 of weeks 1-3. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Dose levels 1-4 must have histologically proven solid malignancy that is metastatic or unresectable with metastatic peritoneal carcinomatosis; as this entity may be difficult to image, peritoneal disease can be documented through other modalities such as operative notes, clinical notes/symptoms, etc as well as imaging
* Dose levels 5 and 6 will be open only to patients with recurrent or persistent primary epithelial ovarian, fallopian or peritoneal cancers; at these dose levels, measurable disease in the abdominal cavity must be present but peritoneal carcinomatosis is not required for eligibility
* Patients must have failed first line standard therapy or have no acceptable standard treatment options; for patients on dose levels 5 and 6, patients may be platinum sensitive, platinum resistant or platinum refractory
* Ability to understand and the willingness to sign a written informed consent document
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Life expectancy of greater than 3 months
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Creatinine =< 1.5 x ULN OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Calcium within normal limit (WNL)
* No surgery, hormonal therapy or chemotherapy within four weeks; for dose levels 5 and 6, patients receiving mitomycin C or nitrosoureas must discontinue treatment 6 weeks prior to registration and any hormonal treatment directed at the malignant tumor must be discontinued at least one week prior to registration; continuation of hormone replacement therapy is permitted
* No previous abdominal radiation; if the patient has received previous pelvic radiation there should not be any overlap between the current and previous radiation fields
* Toxicities of prior chemotherapy recovered to grade 1 or less except for stable grade 2 peripheral neuropathy
* Negative pregnancy test if premenopausal; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Archival tumor sample collection with a tumor block is required for all enrolled patients when available; this will not be required for patients on dose levels 5 and 6; if no block can be released per institutional policy, 10 to 20 unstained slides may be substituted; slides should have a positive charge and a thickness of 3 to 5 microns; if the only tissue sample available is a fine needle aspirate (FNA), the patient will still be considered eligible
* Patients with central nervous system (CNS) metastases to be stable after therapy for > 3 months and off steroid treatment prior to study enrollment
* For patients in dose levels 5 and 6, BRCA testing results, if previously performed, should be attained; if no BRCA testing has been performed, patients may be referred to a genetic counselor and will have detailed family history performed as part of the screening process

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who are currently receiving any other investigational agents
* Brain metastases: patients with treated and stable brain metastasis for 3 months, off steroids will be eligible
* Patients who demonstrate any clinical evidence of bleeding
* Patients who have demonstrated an inability to swallow oral medications
* Patients who currently have an active gastrointestinal obstruction, have had a gastrointestinal obstruction within the last 30 days prior to enrollment and/or are actively requiring parenteral nutrition are excluded; patients who have had a history of any prior gastrointestinal obstruction requiring surgical intervention are also excluded
* Patients who have a known hypersensitivity to the components of the study drug, its analogs or drugs of a similar chemical or biologic composition
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with veliparib
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients who have uncontrolled ascites
* Patients with active seizures or a history of seizure are not eligible
* Patients previously treated with poly (ADP-ribose) polymerase 1 (PARP) inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

PRIMARY OUTCOMES:
Maximum tolerable dose defined as the highest dose at which 0 or 1 dose-limiting toxicities are observed in six patients as graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 28 days
  Reported with exact binomial proportions and 95% confidence intervals.

SECONDARY OUTCOMES:
Changes in quality of life, assessed using the QLQC-30 standardized questionnaire | From baseline to 4 years
  The change in score will be evaluated with a paired t-test. Subscale scores of the quality of life questionnaire will be similarly analyzed.
Clinical activity assessed by response (complete, partial, and overall), measured by RECIST 1.1 criteria | Up to 4 years
  Reported descriptively.
Microsatellite instability (MSI) | Baseline
  MSI will be correlated with response using a Fisher exact test and correlated with progression-free survival (PFS) using the log rank test and Kaplan-Meier curves. The effect of MSI on response and PFS, adjusting for other covariates, will be assessed using logistic regression and the Cox proportional hazards model.
Presence of DNA repair proteins | Baseline
  The presence of ERCC1, XRCC1, BRCA1, BRCA2, and PAR will be categorized by the level of staining: none, mild or strong. These data will be correlated with response and toxicity using the Cochran-Armitage trend test and logistic regression modeling.
Proportion of toxicities of the combination of veliparib and LDRWAR as graded by the NCI CTCAE version 4.0 | Up to 4 weeks after completion of study treatment
  Reported by type and grade with exact binomial proportions and 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (3):
- United States (2):
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada